CLINICAL TRIAL: NCT00292214
Title: Comparative Pharmacokinetics of Intravenous and Oral Paracetamol in the Peri-Operative Period of Laparoscopic Cholecystectomy
Brief Title: Comparing Intravenous and Oral Paracetamol for Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melbourne Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005.138
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2007-03-09 (Estimated); Status verified 2006-02

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: paracetamol; acetaminophen; pharmacokinetic; intravenous; oral; analgesia; pain; opioid
MeSH Terms: conditions — Agnosia; Pain | interventions — Acetaminophen

INTERVENTIONS:
Drug: Paracetamol (acetaminophen)

SUMMARY:
To determine the amount of paracetamol in the blood when given in either intravenous or oral forms prior to cholecystectomy. The clinical effectiveness of each form will also be evaluated with pain scores and the use of other pain relief drugs.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-75
* Scheduled to have elective laparoscopic cholecystectomy under general anaesthesia

Exclusion Criteria:

* Inadequate English comprehension (difficult to obtain informed consent and cooperation), and when interpreters are not available.
* History of allergy or sensitivity to paracetamol
* Administration of oral paracetamol within previous 8 hours
* American Society of Anesthesiologists (ASA) grade IV or V, indicating serious cardio-respiratory co-morbidity
* Not suitable for protocol anaesthetic technique (eg: history of nausea and vomiting with morphine)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-10; Study Completion 2006-10

PRIMARY OUTCOMES:
Early pharmacokinetics (0-240 minutes) of a single dose of 1g paracetamol in IV and oral formulations

SECONDARY OUTCOMES:
Difference in analgesia achieved (15-120 minutes post-operative) with IV and oral paracetamol.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Hogg, Anaesthetist, Principal Investigator — Melbourne Health
Locations (1):
- Royal Melbourne Hospital, Melbourne, Victoria, Australia